CLINICAL TRIAL: NCT02615977
Title: Learning and Decision Making as Predictors of Treatment Outcome in Alcohol Use Disorder (Funding Period 2)
Brief Title: Learning and Relapse Risk in Alcohol Dependence (FP2)
Acronym: LeAD_FP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Charite University, Berlin, Germany (Other); University Hospital Carl Gustav Carus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HE2597/142;ZI1119/32;WI709/102
Record Dates: First submitted 2015-11-20; First posted 2015-11-26 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Alcohol Use Disorder
Keywords: Pavlovian conditioning, Operant conditioning; Pavlovian-to-instrumental transfer; Functional imaging; Relapse risk; Behavioural Intervention
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): In the "verum treatment condition", i.e. Zooming Joystick Task, 90% of all alcohol-related pictures appear in the landscape format and hence are trained to be pushed away.
  Interventions: Behavioral: Zooming Joystick Task
- Placebo Intervention (Placebo Comparator): In the placebo condition, i.e. Zooming Joystick Task (Placebo), alcohol picture are as often pushed away as pulled towards the subject.
  Interventions: Behavioral: Zooming Joystick Task (Placebo)

INTERVENTIONS:
Behavioral: Zooming Joystick Task — Subjects are instructed to use the joystick to pull all pictures (alcoholic and non-alcoholic beverages) towards them that appear in the portrait format, while pictures in a landscape format are pushed away. Half of the pictures are alcohol-related and the other half is not. The assignment of stimuli (alcohol versus neutral) to the picture format (portrait versus landscape) is manipulated (see 'Study Arm' descriptions).
  Arousal and valence of the alcohol and non-alcohol pictures is rated as previously described. The investigators will apply six sessions of ZJT training, as this number has been proven sufficient for reducing relapse rates.
  Other Names: Alcohol Approach Avoidance Task
  Arms: Intervention
Behavioral: Zooming Joystick Task (Placebo) — Subjects are instructed to use the joystick to pull all pictures (alcoholic and non-alcoholic beverages) towards them that appear in the portrait format, while pictures in a landscape format are pushed away. Half of the pictures are alcohol-related and the other half is not. The assignment of stimuli (alcohol versus neutral) to the picture format (portrait versus landscape) is manipulated (see 'Study Arm' descriptions).
  Arousal and valence of the alcohol and non-alcohol pictures is rated as previously described. The investigators will apply six sessions of ZJT training, as this number has been proven sufficient for reducing relapse rates.
  Other Names: Alcohol Approach Avoidance Task (Placebo)
  Arms: Placebo Intervention

SUMMARY:
The investigators will examine clinical alterations in learning and automated approach behaviour and their neurobiological correlates in alcohol-dependent patients and healthy social drinkers and assess whether they are affected by a Zooming Joystick Training (ZJT; randomized "verum" versus "placebo" training) which trains subjects to habitually push alcohol pictures away.

The investigators will test whether activations following treatment predict relapse rate (primary outcome measure) and the prospective amount of alcohol intake (secondary outcome measure) within a six-month follow-up period.

Using fMRI, the investigators will use the Pavlovian-to-Instrumental-Transfer (PIT) paradigm established during the first funding period to distinguish the effects of appetitive, aversive, and drug-related Pavlovian cues on automated instrumental approach behaviour and to assess ZJT training effects comparing functional activation before and after ZJT training.

The investigators will also scan subjects during performance of a short standard working memory task. Behaviourally, aspects of impulsivity will be assessed with the Value-Based Decision Making (VBDM) Battery. Scanning will be repeated after ZJT training to assess its effects on the neural correlates of Pavlovian-to-Instrumental transfer (PIT).

DETAILED DESCRIPTION:
This Project will examine 130 detoxified alcohol-dependent patients and 40 age- and gender matched controls. All subjects will be treated with Zooming Joystick Task (ZJT) training to alter a habitual alcohol cue approach bias. The primary aim of this project is to assess

1. which behavioural and neuroimaging alterations (fMRI) associated with reward-based learning are altered by ZJT treatment and which alterations predict treatment outcome (primary outcome: relapse, secondary outcome: amount of alcohol intake) within the follow-up period of 6 months,
2. how these alterations interact with clinical and psychosocial factors that can modify relapse risk, and
3. to provide data for genetic and imaging analyses and modelling. Furthermore, the investigators will explore gender effects on functional imaging parameters of learning.

Patients will be detoxified in an inpatient setting, receive six sessions of the ZJT in a randomized placebo controlled design and will be followed for six months using the Time-Line Follow-Back Procedure. Clinical assessments, behavioural paradigms of learning, and brain imaging will be carried out within at least four half-lives after any psychotropic medication. Subjects will undergo medical management with biweekly follow-ups and predefined inclusion and exclusion criteria as previously described. Functional imaging paradigms will be applied, assessing

1. Pavlovian-to-instrumental transfer,
2. habitual versus goal directed behaviour and
3. working memory.

The investigators will associate model parameters of learning with functional activation and prospective intake controlling for comorbidity, psychosocial and neurobiological disease severity markers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-65 years
* alcohol dependence/alcohol use disorder according to ICD-10 and alcohol-use disorder according to DSM-5
* Minimum of 72 hours of abstinence, maximum of 21 days of abstinence
* Minimum of three years with alcohol dependence/alcohol use disorder
* Low severity of withdrawal symptoms
* Ability to provide fully informed consent and to use self-rating scales
* Sufficient understanding of the German language

Exclusion Criteria:

* Lifetime history of DSM-IV bipolar, psychotic disorder, or substance dependence other than nicotine dependence. Patients may have had lifetime alcohol dependence/alcohol use disorder diagnoses.
* Current threshold DSM-IV diagnosis of any of the following disorders: current (hypo)manic episode, major depressive disorder, generalized anxiety disorder, PTSD, borderline personality disorder, or obsessive compulsive disorder
* History of substance dependence other than alcohol or nicotine dependence
* Current substance use other than nicotine and alcohol as evinced by positive urine test
* History of severe head trauma or other severe central neurological disorder (dementia, Parkinson's disease, multiple sclerosis)
* Pregnancy or nursing infants
* Any alcohol intake within the last 24 hours
* Use of medications or drugs known to interact with the central nervous system within the last 10 days, except detoxification treatment with benzodiazepines or clomethiazole, with testing at least four half-lives post last intake

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
relapse to heavy drinking | 6 months
  defined as the consumption of over 60g of alcohol per occasion in men and of over 40g of alcohol in women

SECONDARY OUTCOMES:
amount of alcohol intake during the follow-up period | 6 months
  Timeline Followback interview for each day during the follow-up period
blood oxygenation level-dependent (BOLD) signal | at assessment and after last training (approx. 2 weeks after assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Heinz, Prof PhD MD, Study Chair — Charite University, Berlin, Germany; Hans-Ulrich Wittchen, Prof PhD, Study Director — Technische Universität Dresden, Dresden, Germany
Locations (3):
- Germany (3):
  - Universitaetsklinikum Carl Gustav Carus at the Technische Universitaet Dresden, Dresden, Saxony
  - Charité - Universitätsmedizin Berlin, Berlin
  - Technische Universität Dresden, Dresden

REFERENCES:
- [Derived] Zindler T, Frieling H, Fliedner L, Veer IM, Neyazi A, Awasthi S, Ripke S, Walter H, Friedel E. How alcohol makes the epigenetic clock tick faster and the clock reversing effect of abstinence. Addict Biol. 2022 Sep;27(5):e13198. doi: 10.1111/adb.13198. PMID 36001430
- See also: English study description — http://gepris.dfg.de/gepris/projekt/186318919?language=en